CLINICAL TRIAL: NCT03612544
Title: Substudy of Efficacy, Safety and Toxicology of Electronic Nicotine Delivery Systems as an Aid for Smoking Cessation (ESTxENDS Trial)- the Toxins Substudy of ESTxENDS
Brief Title: The ESTxENDS Trial- Substudy on the Effect on Toxins From Using Electronic Nicotine Delivery Systems (ENDS/Vaporizer/E-cig)
Acronym: ESTxENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Lausanne (Other); University of Geneva, Switzerland (Other); University of Zurich (Other); State Hospital, St. Gallen (Other Government); Swiss National Science Foundation (Other); Krebsforschung Schweiz, Bern, Switzerland (Other); Federal Office of Public Health, Switzerland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-02332e
Record Dates: First submitted 2018-07-02; First posted 2018-08-02 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; Toxicity
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Masking Description: Statisticians and laboratory personnel will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: ENDS (Vaporizer/e-cig) and smoking cessation counseling
- Control group (Active Comparator)
  Interventions: Other: Smoking cessation counseling

INTERVENTIONS:
Other: ENDS (Vaporizer/e-cig) and smoking cessation counseling — Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Intervention group
Other: Smoking cessation counseling — Participants in the control group will receive smoking cessation counseling only. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Control group

SUMMARY:
--> This is a substudy of the main ESTxENDS trial (NCT03589989). Toxins outcomes should be considered secondary outcomes of the main smoking cessation outcome formulated in NCT03589989.

Cigarette smoking is the leading cause of preventable death in Switzerland. Recently, electronic nicotine delivery systems (ENDS; also called vaporizer or electronic cigarette) have become popular with smokers who want to stop smoking or reduce their exposure to inhaled chemicals since ENDS use appears to be safer than tobacco smoking.

Conventional cigarettes release toxic chemicals in tobacco smoke through thermochemical degradation and pyrolysis processes by combusting tobacco, but in ENDS toxicants can be released by heating up nicotine-containing e-liquids to produce vapor. The e-liquid in ENDS is mostly made of propylene glycol (PG) and vegetal glycerin (VG) in addition to nicotine, flavorings and sometimes alcohol as a conservation agent. The heating process of the e-liquid in ENDS, has been shown to release carcinogens such as some carbonyl and volatile organic compounds (i.e., formaldehyde, acetaldehyde and acrolein). Some devices might also release heavy metals such as cadmium, lead and mercury. The source of such metals may be the metal of the device or the e-liquids. Although unexpected from the composition of the e-liquids, some studies have also detected tobacco-specific nitrosamines (TNSAs) (N'-nitrosonornicotine (NNN) and 4-(methylnitrosoamino)-1-(3-pyridyl)-1-butanone (NNK)) and polycyclic aromatic hydrocarbons (PAHs) (1- and 2-Naphtol and 1-hydroxypyrene (1-OHP)).

This study will therefore test the efficacy of ENDS for cigarette smoking cessation, the safety of ENDS on adverse events and the effect of ENDS on health-related outcomes and exposure to inhaled chemicals.

For the main ESTxENDS trial (NCT03589989), cigarette smokers motivated to quit smoking cigarettes will be included. Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants in the control group will receive smoking cessation counseling only. All participants will be followed over a 24-month period. Chemicals such as VOCs, PAHs, TSNAs, heavy metals, nicotine and nicotine degradation products will first be quantified in the aerosol produced by ENDS in laboratory conditions. These chemicals and their metabolites will then be measured at baseline and at 6-, 12- and 24- months' follow-up in urine samples from study participants.

ELIGIBILITY:
Inclusion criteria:

* Informed Consent as documented by signature
* Persons aged 18 or older
* Currently smoking 5 or more cigarettes a day for at least 12 months
* Willing to try to quit smoking within the next 3 months,
* Persons providing a valid phone number, a valid email address and/or a valid postal address.

Exclusion criteria:

* Known hypersensitivity or allergy to contents of the e-liquid
* Participation in another study with investigational drug within the 30 days preceding the baseline visit and during the present study where interactions are to be expected
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the scheduled study intervention, i.e. within the first 6-months of the study
* Persons having used ENDS or tobacco heating systems regularly in the 3 months preceding the baseline visit
* Persons having used nicotine replacement therapy (NRT) or other medications with demonstrated efficacy as an aid for smoking cessation such as varenicline or bupropion within the 3 months preceding the baseline visit
* Persons who cannot attend the 6- month follow-up visit for any reason
* Cannot understand instructions delivered in person or by phone, or otherwise unable to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Concentrations of urinary NNAL (4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol)_1 | 6 months post quit date
  Measurement of NNAL (4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol) in urine
Concentrations of urinary NNAL (4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol)_2 | 12 months post quit date
  Measurement of NNAL (4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol) in urine
Concentrations of urinary NNAL (4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol)_3 | 24 months post quit date
  Measurement of NNAL (4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol) in urine
Concentrations of urinary NNN (N-nitrosonornicotine)_1 | 6 months post quit date
  Measurement of NNN (N-nitrosonornicotine) in urine
Concentrations of urinary NNN (N-nitrosonornicotine)_2 | 12 months post quit date
  Measurement of NNN (N-nitrosonornicotine) in urine
Concentrations of urinary NNN (N-nitrosonornicotine)_3 | 24 months post quit date
  Measurement of NNN (N-nitrosonornicotine) in urine
Concentrations of urinary NNK (nicotine-derived nitrosamine ketone)_1 | 6 months post quit date
  Measurement of NNK (nicotine-derived nitrosamine ketone) in urine
Concentrations of urinary NNK (nicotine-derived nitrosamine ketone)_2 | 12 months post quit date
  Measurement of NNK (nicotine-derived nitrosamine ketone) in urine
Concentrations of urinary NNK (nicotine-derived nitrosamine ketone)_3 | 24 months post quit date
  Measurement of NNK (nicotine-derived nitrosamine ketone) in urine
Concentrations of urinary metabolites of VOCs (volatile organic compounds)_1 | 6 months post quit date
  Measurements of metabolites of VOCs in urine
Concentrations of urinary metabolites of VOCs (volatile organic compounds)_2 | 12 months post quit date
  Measurements of metabolites of VOCs in urine
Concentrations of urinary metabolites of VOCs (volatile organic compounds)_3 | 24 months post quit date
  Measurements of metabolites of VOCs in urine
Concentrations of urinary PAHs (Polycyclic aromatic hydrocarbons)_1 | 6 months post quit date
  Measurement of PAHs (Polycyclic aromatic hydrocarbons) in urine
Concentrations of urinary PAHs (Polycyclic aromatic hydrocarbons)_2 | 12 months post quit date
  Measurement of PAHs (Polycyclic aromatic hydrocarbons) in urine
Concentrations of urinary PAHs (Polycyclic aromatic hydrocarbons)_3 | 24 months post quit date
  Measurement of PAHs (Polycyclic aromatic hydrocarbons) in urine
Concentrations of urinary heavy metals_1 | 6 months post quit date
  Measurement of heavy metals in urine
Concentrations of urinary heavy metals_2 | 12 months post quit date
  Measurement of heavy metals in urine
Concentrations of urinary heavy metals_3 | 24 months post quit date
  Measurement of heavy metals in urine
Concentrations of urinary nicotine metabolites_1 | 6 months post quit date
  Measurement of nicotine metabolites in urine
Concentrations of urinary nicotine metabolites_2 | 12 months post quit date
  Measurement of nicotine metabolites in urine
Concentrations of urinary nicotine metabolites_3 | 24 months post quit date
  Measurement of nicotine metabolites in urine

SECONDARY OUTCOMES:
Change in concentrations of urinary NNAL (4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol) | Change from baseline to 6,12, 24 months post quit date
  Change of NNAL (4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol) concentrations in urine from baseline to 6, 12, and 24 months post quit date.
Change in concentrations of urinary NNN (N-nitrosonornicotine) | Change from baseline to 6,12, 24 months post quit date
  Change of NNN (N-nitrosonornicotine) concentrations in urine from baseline to 6, 12, and 24 months post quit date.
Change in concentrations of urinary NNK (nicotine-derived nitrosamine ketone) | Change from baseline to 6,12, 24 months post quit date
  Change of NNK (nicotine-derived nitrosamine ketone) concentrations in urine from baseline to 6, 12, and 24 months post quit date.
Change in concentrations of urinary VOCs (volatile organic compounds) | Change from baseline to 6,12, 24 months post quit date
  Change of VOCs (volatile organic compounds) concentrations in urine from baseline to 6, 12, and 24 months post quit date.
Change in concentrations of urinary PAHs (Polycyclic aromatic hydrocarbons) | Change from baseline to 6,12, 24 months post quit date
  Change of PAHs (Polycyclic aromatic hydrocarbons) concentrations in urine from baseline to 6, 12, and 24 months post quit date.
Change in concentrations of urinary heavy metals | Change from baseline to 6,12, 24 months post quit date
  Change of heavy metals concentrations in urine from baseline to 6, 12, and 24 months post quit date.
Change in concentrations of urinary nicotine metabolites | Change from baseline to 6,12, 24 months post quit date
  Change of nicotine metabolites concentrations in urine from baseline to 6, 12, and 24 months post quit date.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, Prof.Dr.med, Study Director — Berner Institut für Hausarztmedizin; Universität Bern
Locations (5):
- Switzerland (5):
  - Unisanté, Centre universitaire de médecine générale et santé publique, Université de Lausanne, Lausanne, Canton of Vaud
  - University Clinic for General Internal Medicine, Bern University Hospital, Bern
  - Département de médecine interne, Hôpitaux universitaires de Genève, Geneva
  - Lungenzentrum, Klinik für Pneumologie und Schlafmedizin, Kantonsspital St. Gallen, Sankt Gallen
  - Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich, Zurich

REFERENCES:
- [Background] Farsalinos KE, Polosa R. Safety evaluation and risk assessment of electronic cigarettes as tobacco cigarette substitutes: a systematic review. Ther Adv Drug Saf. 2014 Apr;5(2):67-86. doi: 10.1177/2042098614524430. PMID 25083263
- [Background] Orr MS. Electronic cigarettes in the USA: a summary of available toxicology data and suggestions for the future. Tob Control. 2014 May;23 Suppl 2(Suppl 2):ii18-22. doi: 10.1136/tobaccocontrol-2013-051474. PMID 24732158
- [Background] Bertholon JF, Becquemin MH, Roy M, Roy F, Ledur D, Annesi Maesano I, Dautzenberg B. [Comparison of the aerosol produced by electronic cigarettes with conventional cigarettes and the shisha]. Rev Mal Respir. 2013 Nov;30(9):752-7. doi: 10.1016/j.rmr.2013.03.003. Epub 2013 Apr 17. French. PMID 24267765
- [Background] Etter JF, Bullen C. Electronic cigarette: users profile, utilization, satisfaction and perceived efficacy. Addiction. 2011 Nov;106(11):2017-28. doi: 10.1111/j.1360-0443.2011.03505.x. Epub 2011 Jul 27. PMID 21592253
- [Background] Etter JF, Zather E, Svensson S. Analysis of refill liquids for electronic cigarettes. Addiction. 2013 Sep;108(9):1671-9. doi: 10.1111/add.12235. Epub 2013 May 23. PMID 23701634
- [Background] Flouris AD, Poulianiti KP, Chorti MS, Jamurtas AZ, Kouretas D, Owolabi EO, Tzatzarakis MN, Tsatsakis AM, Koutedakis Y. Acute effects of electronic and tobacco cigarette smoking on complete blood count. Food Chem Toxicol. 2012 Oct;50(10):3600-3. doi: 10.1016/j.fct.2012.07.025. Epub 2012 Jul 31. PMID 22858449
- [Background] Goniewicz ML, Knysak J, Gawron M, Kosmider L, Sobczak A, Kurek J, Prokopowicz A, Jablonska-Czapla M, Rosik-Dulewska C, Havel C, Jacob P 3rd, Benowitz N. Levels of selected carcinogens and toxicants in vapour from electronic cigarettes. Tob Control. 2014 Mar;23(2):133-9. doi: 10.1136/tobaccocontrol-2012-050859. Epub 2013 Mar 6. PMID 23467656
- [Background] Ingebrethsen BJ, Cole SK, Alderman SL. Electronic cigarette aerosol particle size distribution measurements. Inhal Toxicol. 2012 Dec;24(14):976-84. doi: 10.3109/08958378.2012.744781. PMID 23216158
- [Background] McAuley TR, Hopke PK, Zhao J, Babaian S. Comparison of the effects of e-cigarette vapor and cigarette smoke on indoor air quality. Inhal Toxicol. 2012 Oct;24(12):850-7. doi: 10.3109/08958378.2012.724728. PMID 23033998
- [Background] Pellegrino RM, Tinghino B, Mangiaracina G, Marani A, Vitali M, Protano C, Osborn JF, Cattaruzza MS. Electronic cigarettes: an evaluation of exposure to chemicals and fine particulate matter (PM). Ann Ig. 2012 Jul-Aug;24(4):279-88. PMID 22913171
- [Background] Uchiyama S, Ohta K, Inaba Y, Kunugita N. Determination of carbonyl compounds generated from the E-cigarette using coupled silica cartridges impregnated with hydroquinone and 2,4-dinitrophenylhydrazine, followed by high-performance liquid chromatography. Anal Sci. 2013;29(12):1219-22. doi: 10.2116/analsci.29.1219. PMID 24334991
- [Background] Walton KM, Abrams DB, Bailey WC, Clark D, Connolly GN, Djordjevic MV, Eissenberg TE, Fiore MC, Goniewicz ML, Haverkos L, Hecht SS, Henningfield JE, Hughes JR, Oncken CA, Postow L, Rose JE, Wanke KL, Yang L, Hatsukami DK. NIH electronic cigarette workshop: developing a research agenda. Nicotine Tob Res. 2015 Feb;17(2):259-69. doi: 10.1093/ntr/ntu214. Epub 2014 Oct 21. PMID 25335949